CLINICAL TRIAL: NCT01939457
Title: Introduction of 400mcg Sublingual Misoprostol as First Line Treatment in 11 Health Posts in Three Districts in Senegal
Brief Title: 400mcg Sublingual Misoprostol as First Line Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2.2.4
Record Dates: First submitted 2013-08-07; First posted 2013-09-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Incomplete Abortion
MeSH Terms: conditions — Abortion, Incomplete | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- misoprostol (Experimental): 400 mcg misoprostol sublingually
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol

SUMMARY:
Women presenting with incomplete abortion and eligible for treatment with misoprostol were offered 400mcg sublingual misoprostol for treatment. Based on existing literature, the study hypothesises that women can successfully be treated with misoprostol alone as first line treatment.

ELIGIBILITY:
Inclusion Criteria:

* uterine size less than 12 weeks lmp
* open cervical os
* current or past vaginal bleeding
* willing to provide contact information for follow-up
* over 18 or with guardian consent

Exclusion Criteria:

* suspicion of ectopic pregnancy
* intrauterine device in place
* bad general health (infection, anemia, shoc)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2011-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
complete abortion | 1 year
  number of complete abortion with misoprostol treatment alone

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD MPH, Principal Investigator — Gynuity Health Projects
Locations (1):
- Guediawaye Health Center, Guédiawaye, Senegal

REFERENCES:
- [Derived] Gaye A, Diop A, Shochet T, Winikoff B. Decentralizing postabortion care in Senegal with misoprostol for incomplete abortion. Int J Gynaecol Obstet. 2014 Sep;126(3):223-6. doi: 10.1016/j.ijgo.2014.03.028. Epub 2014 May 15. PMID 24893962